CLINICAL TRIAL: NCT06257979
Title: Unexpected Positive Cultures in Rotator Cuff Revision Surgery: Significance and Influence on Outcomes and Tendon Healing
Brief Title: Unexpected Positive Cultures in Rotator Cuff Revision Surgery
Acronym: POCICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-A02042-43
Record Dates: First submitted 2024-01-05; First posted 2024-02-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Rotator Cuff Repair
Keywords: Unexpected Positive Cultures (UPC); Revision cuff repair surgery (RCR)

STUDY DESIGN:
Intervention Model Description: The study procedure involves a re-intervention of the rotator cuff, which is conducted for the patients in accordance with standard practice. The patient undergoes local and/or general anesthesia, along with intravenous or oral antibiotic prophylaxis.
  During the intervention, the surgeon collects the sutures placed during the first intervention, the product of tendon debridement, and the subacromial bursa (cleaning product) used during the re-intervention. These elements usually discarded, are collected for the bacteriological analysis.
  Antibiotic treatment cannot be prescribed immediately and during the first month following this re-intervention (time for biofilm formation). As per the protocol, even a positive sample should not lead to the initiation of systematic antibiotic therapy. In the case of identification of a pathogenic microorganism, antibiotic therapy will be prescribed, leading to discontinuation of the study.
Who Masked: Participant
Masking Description: Following the analysis of the bacteriological samples, the investigator will read the bacteriological results. These will be entered into the database.
  During subsequent visits, the investigator will not provide this information to the patient who will thus remain as a single blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Other): Operated patients with positive results for their pre-operative microbiological samples.
  Interventions: Other: This study is with minimal risk and minimal constraints due to the addition of questionnaires
- Control group (Other): Operated patients with negative results for their pre-operative microbiological samples.
  Interventions: Other: This study is with minimal risk and minimal constraints due to the addition of questionnaires

INTERVENTIONS:
Other: This study is with minimal risk and minimal constraints due to the addition of questionnaires — In this study, the specific procedures compared to routine care are :
  * Considering the addition of questionnaires, this study will be prospective. Due to the use of bacteriological samples, it is considered as a minimal-risk research.
  * The research procedure involves a bacteriological analysis of operative elements (sutures placed during the first intervention, the product of tendon debridement, and the subacromial bursa (cleaning product)) used during the re-intervention. These usually discarded operative samples are collected for bacteriological analysis.
  * Antibiotic treatment cannot be prescribed immediately after the surgery and during the first month following this re-intervention (time for biofilm formation). As per the protocol, even a positive sample should not lead to the initiation of systematic antibiotic therapy. In the case of identification of a pathogenic microorganism, antibiotic therapy will be prescribed, leading to discontinuation of the study.
  Other Names: Microbiological analysis of samples collected from operated patients: in the presence of UPC, it does not influence the postoperative course; No antibiotics are prescribed during the first month after the operation.

SUMMARY:
In the context of rotator cuff re-intervention, the impact of Unexpected Positive Cultures (UPC) is not documented, and their management has not been studied, particularly regarding indications for antibiotic therapy, which is currently not a consensus.

A prospective interventional study will be implemented to compare the results of non-randomized patient samples, whether positive or negative, taken during rotator cuff re-intervention. The objective is to assess whether these samples do not affect clinical outcomes and tendon healing rates.

DETAILED DESCRIPTION:
Rotator cuff injuries are a common pathology with a 30% prevalence in the general population. If rotator cuff repair fails, patients often experience persistent pain, and bacteria can be detected during the revision period in approximately 30% of cases, even in the absence of septic symptoms. This type of infection, referred to as low-level infection, occurs in around 5% of cases and is frequently implicated as a contributing factor to poor outcomes of the intervention.

Bacteriological samples are routinely collected during revisions, especially for prostheses. The appropriate course of action in cases where these samples test positive, yet there are no signs of infection, remains to be clarified. Notably, administering antibiotics in response to unexpected positive cultures (UPC) during the revision period for total shoulder prostheses does not appear to significantly impact results or infection rates.

In the context of rotator cuff re-interventions, the impact of UPC has not been well-documented. The management of UPC, particularly regarding antibiotic therapy, has not been thoroughly studied and is not currently recommended. Further research is needed to establish guidelines for managing positive cultures in the absence of infection symptoms during rotator cuff re-interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 or over
* Patient requiring re- intervention for Rotator Ruff Revision Surgery for non-healing of the same tendons after a first intervention (delay <2 years)
* Patient requiring arthroscopy
* Patient having had realized a MRI of the shoulder in the 6 previous months
* Affiliate participant or beneficiary of a social security scheme
* Participant having been informed and not having objected to the use of their data

Exclusion Criteria:

* Patient with at least one clinical sign of infection (fever, redness)
* Patient with a new distant rupture on a healed cuff (> 3 years)
* Patient with a history of shoulder surgery other than initial Rotator Ruff Surgery
* Patient having received antibiotic treatment in the 2 weeks preceding inclusion
* Participant in another research
* Participant in a period of exclusion from another research still in progress at the time of inclusion
* Protected participant: an adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Participant hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Compare the functional recovery of the shoulder at one year after iterative repair of non-healing rotator cuff between patients with unexpected positive cultures and patients with negative results. | at Month 1, Month 3, Month 6 and 1 Year after the re-intervention
  Compare the functional recovery (Yes/No), at one year after iterative repair of non-healing rotator cuff between patients with unexpected positive cultures and patients with negative results using the Constant Score.
Compare the 2 groups on tendon healing, after iterative repair of non-healing of the rotator cuff | at Month 1, Month 3, Month 6 and 1 Year after the re-intervention
  Compare the 2 groups on tendon healing (Yes/No), after iterative repair of non-healing of the rotator cuff using the Constant Score.
Compare the 2 groups on the occurrence of post-operative complications, after iterative repair of non-healing of the rotator cuff | up to one year after the re-intervention
  Compare the 2 groups on the occurrence of post-operative complications (Yes/No), after iterative repair of non-healing of the rotator cuff and list them
Compare the 2 groups on the patient's other functional scores | at Month 1, Month 3, Month 6 and 1 Year after the re-intervention
  Compare the 2 groups on the patient's other functional scores such as SSV and ASES questionnaries
Describe the pathogenic germs found in the positive cultures | at Month 1 after the re-intervention
  List of pathogenic germs found in the positive samples

SECONDARY OUTCOMES:
Sugaya score measured from MRI to assess the influence of positive cultures on tendon healing | at one year after the re-intervention
  The quality of the repair was assessed using an MRI and the Sugaya classification (French version):
  Type 1: Normal thickness and echostructure of the rotator cuff. Type 2: Normal thickness and heterogeneous echostructure. Type 3: Thinning without discontinuity. Type 4: Moderate discontinuity. Type 5: Frank discontinuity.
Occurrence of complications during the first post-operative year | up to one year after the re-intervention
  List of of complications during the first post-operative year
Functional scores at one year: American Shoulder and Elbow Surgeons Score (ASES) | at one year after the re-intervention
  ASES score can be viewed as a 100-point scale that evaluates two dimensions of shoulder function: pain and performance in activities of daily living. Each of the two domains make up for 50 of the 100 points.
Functional scores at one year: Subjective Shoulder Value (SSV) | at one year after the re-intervention
  SSV score is defined as the subjective evaluation by the patient of shoulder function, expressed as a percentage of a normal shoulder. This score ranges from 0 to 100%.
Pathogenic bacteria detected in the group of patients with positive results | at Month 1 after the re-intervention
  List of pathogenic bacteria detected in the group of patients with positive results

CONTACTS AND LOCATIONS:
Overall Officials: Maxime ANTONI, MD, Study Director — Clinique de l'Orangerie-Strasbourg
Locations (8):
- France (8):
  - Hôpital privé La Châtaigneraie ELSAN, Beaumont
  - Hôpital privé Saint-Martin, Caen
  - Clinique Louis Pasteur, Essey-lès-Nancy
  - Santy-Lyon-Ramsay, Lyon
  - Clinique d'occitanie ELSAN, Muret
  - ICR-Kantys, Nice
  - Santé Atlantique ELSAN, Saint-Herblain
  - Clinique de l'Orangerie, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao J, Luo M, Pan J, Liang G, Feng W, Zeng L, Yang W, Liu J. Risk factors affecting rotator cuff retear after arthroscopic repair: a meta-analysis and systematic review. J Shoulder Elbow Surg. 2021 Nov;30(11):2660-2670. doi: 10.1016/j.jse.2021.05.010. Epub 2021 Jun 2. PMID 34089878
- [Background] Azar M, Van der Meijden O, Pireau N, Chelli M, Gonzalez JF, Boileau P. Arthroscopic revision cuff repair: do tendons have a second chance to heal? J Shoulder Elbow Surg. 2022 Dec;31(12):2521-2531. doi: 10.1016/j.jse.2022.04.024. Epub 2022 Jun 6. PMID 35671929
- [Background] Bonnevialle N, Dauzeres F, Toulemonde J, Elia F, Laffosse JM, Mansat P. Periprosthetic shoulder infection: an overview. EFORT Open Rev. 2017 Apr 27;2(4):104-109. doi: 10.1302/2058-5241.2.160023. eCollection 2017 Apr. PMID 28507783
- [Background] Neufeld ME, Lanting BA, Shehata M, Naudie DDR, McCalden RW, Teeter MG, Vasarhelyi EM. The Prevalence and Outcomes of Unexpected Positive Intraoperative Cultures in Presumed Aseptic Revision Knee Arthroplasty. J Arthroplasty. 2022 Nov;37(11):2262-2271. doi: 10.1016/j.arth.2022.05.036. Epub 2022 May 19. PMID 35598759
- [Background] Falstie-Jensen T, Lange J, Daugaard H, Sorensen AKB, Ovesen J, Soballe K; ROSA Study Group. Unexpected positive cultures after revision shoulder arthroplasty: does it affect outcome? J Shoulder Elbow Surg. 2021 Jun;30(6):1299-1308. doi: 10.1016/j.jse.2020.12.014. Epub 2021 Feb 3. PMID 33548396
- [Background] Hodakowski AJ, Cohn MR, Mehta N, Menendez ME, McCormick JR, Garrigues GE. An evidence-based approach to managing unexpected positive cultures in shoulder arthroplasty. J Shoulder Elbow Surg. 2022 Oct;31(10):2176-2186. doi: 10.1016/j.jse.2022.03.019. Epub 2022 May 2. PMID 35513254
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Sugaya H, Maeda K, Matsuki K, Moriishi J. Functional and structural outcome after arthroscopic full-thickness rotator cuff repair: single-row versus dual-row fixation. Arthroscopy. 2005 Nov;21(11):1307-16. doi: 10.1016/j.arthro.2005.08.011. PMID 16325080
- [Background] Angst F, Goldhahn J, Drerup S, Aeschlimann A, Schwyzer HK, Simmen BR. Responsiveness of six outcome assessment instruments in total shoulder arthroplasty. Arthritis Rheum. 2008 Mar 15;59(3):391-8. doi: 10.1002/art.23318. PMID 18311752
- [Background] Gilbart MK, Gerber C. Comparison of the subjective shoulder value and the Constant score. J Shoulder Elbow Surg. 2007 Nov-Dec;16(6):717-21. doi: 10.1016/j.jse.2007.02.123. PMID 18061114